CLINICAL TRIAL: NCT01111084
Title: Prospective Multi-centre Observational Study to Determine the Mono-bifollicular Development in Infertile Women Subjected to Ovulation Induction With Follitropin α
Brief Title: A Prospective, Multi-centric Observational Study to Determine the Mono-bifollicular Development in Infertile Women Subjected to Ovulation Induction With Follitropin α
Acronym: P450
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Dr. Sebastián Burgués/Medical Manager, Merck Serono Spain, an affilaite of MerckKGaA, Darmstadt, Germany
Other Study IDs: IMP24846
Record Dates: First submitted 2010-04-23; First posted 2010-04-27 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2010-04

CONDITIONS: Ovulation Induction
Keywords: Ovulation induction; Ovarian Hyperstimulation Syndrome; Pregnancy; Fertility
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome | interventions — Glycoprotein Hormones, alpha Subunit; follitropin alfa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum

INTERVENTIONS:
Drug: Follitropin alpha (r-FSH) — The dosage and administration of follitropin alpha was according to each centre's protocol and within technical specification recommendations.
  Other Names: Gonal-f

SUMMARY:
This is a prospective and multicentric observational study to determine the real mono-bifollicular development rate that is obtained under normal care conditions following ovulation induction (OI) treatment with follitropin-alpha filled by mass prescribed in accordance with standard practice.

DETAILED DESCRIPTION:
In women with infertility due to anovulation, the main purpose of ovulation induction (OI) consists in inducing the mono or bifollicular and the subsequent ovulation in order to achieve pregnancy. The availability of recombinant gonadotropins obtained using genetically engineered techniques has meant a decisive and clear pharmacological advancement. Use of recombinant human follicle stimulating hormone (r-hFSH) offers a greater effectiveness (greater number of follicles/ ovocytes and a higher pregnancy rate) and efficiency (fewer number of blisters, fewer stimulation days; fewer number of cancellations and complications) in programmed coitus and artificial insemination like in-vitro fertilisation (IVF)/intra cytoplasmic sperm injection (ICSI) techniques. Further advances in obtaining better products for ovarian stimulation has led to production of a recombinant FSH (follitropin alpha) filled by mass preparation. This hormone becomes the most consistent and precise gonadotropin due to improvements in its quantification process.

Today, despite having accurate and modern tools for ovulation induction, in daily practice, doctors continue to "fight" against two old problems of assisted reproduction: multiple pregnancies and ovarian hyperstimulation syndrome (OHSS). Application of assisted reproduction techniques (ARTs) and the use of medication that induce ovulation, risk producing gestations and multiple births with a higher frequency than those observed in spontaneous gestations. One of the facts that result in the appearance of such problems is the high incidence of polycystic ovarian syndrome among the population of women who are infertile due to anovulation. These subjects are especially sensitive to ovarian stimulation, which leads to multiple follicular development, a higher risk of hyperstimulation and higher rates of multiple pregnancies.

Therefore, it seems clear that the search for developing mono or bifollicular cycles is important in ovarian induction cycles, for the purpose of preventing the above mentioned multiple pregnancy problems and the risk of OHSS. The intent of this study was to figure out the real mono-bifollicular development rate that is obtained under normal care conditions following OI treatment with follitropin alpha filled by mass prescribed in accordance with standard practice. Therefore, a measure of the efficiency of the product for achieving the development of one or two follicles. Data was collected from 56 centres of the Autonomous Communities that accepted this observational study, until achieving a total of 410 ovulation induction cycles.

OBJECTIVES

Primary objective:

* To find the real proportion of cycles with mono-bifollicular development during the provision of care involving OI with follitropin alpha filled by mass

Secondary objectives:

* To evaluate if the use of follitropin alpha filled by mass has other clinical benefits such as a reduction in the number of cancelled cycles, of the dosage and time required and adverse effects

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women with infertility caused by anovulation, who wished to conceive and were included in an ovulation induction (OI) treatment protocol for intrauterine insemination or for programmed coitus

Exclusion Criteria:

* Subjects with hypersensitivity to follitropin alpha, to FSH or to any of the excipients
* Subjects with hypothalamic or pituitary tumours
* Subjects with increase in the size of the ovaries or cysts that were not due to polycystic ovary disease
* Subjects with gynaecologic haemorrhages of unknown aetiology
* Subjects with ovarian, uterine or mammary carcinoma
* Subjects with primary ovarian failure
* Subjects with malformations of sex organs that were not compatible with pregnancy
* Subjects with uterine fibroid tumours that were not compatible with pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female subjects who were infertile due to anovulation undergoing OI treatment with follitropin alpha prescribed in accordance with the standard practice and in accordance with the technical specifications.
Sampling Method: Non-Probability Sample
Enrollment: 410 (Actual)
Dates: Start 2004-03; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Follicular development | First 10 months from the inclusion of the subjects
  Number and size of follicles as determined through transvaginal ultrasound

SECONDARY OUTCOMES:
Secondary efficacy assessments | From baseline until the pregnancy or menstruation confirmation
  Duration of ovulation induction; total accumulated dosage of follitropin alpha; cycles cancelled due to insufficient response or due to risk of ovarian hyperstimulation; proportion of pregnancies
Safety assessments | First 10 months from the inclusion of the subjects
  Incidence of adverse occurrences, in particular OHSS; proportion of multiple pregnancies and local reaction at the injection point.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Enrique Granados, Study Director — Merck Serono Spain
Locations (1):
- Hospital Ntra. Sra. De Valme, Seville, Spain